CLINICAL TRIAL: NCT00001665
Title: Can Subthreshold Transcranial Magnetic Stimulation (rTMS) to Motor Cortex and/or to Supplementary Motor Area (SMA) Improve Performance of Complex Motor Sequences in Parkinson's Disease?
Brief Title: Transcranial Magnetic Stimulation for the Treatment of Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970073; 97-N-0073
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-12

CONDITIONS: Movement Disorders; Parkinson Disease
Keywords: Magnetic Stimulation; Motor Skills; Parkinson's Disease; rTMS
MeSH Terms: conditions — Movement Disorders; Parkinson Disease

SUMMARY:
The problems in motor activity associated with Parkinson's disease are still poorly understood. Patients with Parkinson's disease often suffer from extremely slow movements (bradykinesia) which result in the inability to perform complex physical acts.

Imaging studies of the brain have provided researchers with information about the specific areas in the brain associated with these motor difficulties. One particular area involved is the surface of the brain called the cerebral cortex.

Transcranial Magnetic Stimulation (TMS) is a non-invasive technique that can be used to stimulate brain activity and gather information about brain function. It is very useful when studying the areas of the brain related to motor activity (motor cortex, corticospinal tract, and corpus callosum). Repetitive transcranial magnetic stimulation (rTMS) involves the placement of a cooled electromagnet with a figure-eight coil on the patient's scalp and rapidly turning on and off the magnetic flux. This permits non-invasive, relatively localized stimulation of the surface of the brain (cerebral cortex). The effect of magnetic stimulation varies, depending upon the location, intensity and frequency of the magnetic pulses.

Researchers plan to study the therapeutic effects of repetitive transcranial magnetic stimulation (rTMS) on complex motor behavior of patients with Parkinson's disease. In order to measure its effectiveness, patients will be asked to perform complex tasks, such as playing the piano while receiving transcranial magnetic stimulation.

DETAILED DESCRIPTION:
The physiology of the motor disturbance in Parkinson's disease is not completely understood. One of the major and perhaps most disabling manifestations of PD is bradykinesia. It is particularly difficult for these patients to perform simultaneous, sequential and complex motor acts. Imaging studies have recently provided important information in reference to the brain regions associated with performance of these motor sequences in normal volunteers and in PD patients. These studies helped us to identify the brain regions active in association with task performance. It has been suggested that cortical regions, and particularly the SMA are less active in patients with PD than in controls in association with motor performance.

We plan to study the effects of subthreshold rTMS delivered to SMA and primary motor cortex in patients with PD "on" and "off" medication. From this study, we expect to learn if stimulation of the scalp overlying primary motor cortex and SMA can ameliorate performance of simple and complex motor sequences in PD.

Subthreshold rTMS has been proposed as a therapeutic tool in psychiatric disorders. In the motor domain, subthreshold rTMS delivered to primary motor cortex improves reaction times and motor performance in patients with Parkinson's disease. The mechanisms underlying this beneficial effect are not known. However, they may be related with subthreshold rTMS replacing the missing excitatory drive on the motor cortex.

ELIGIBILITY:
Patients with PD.

No epilepsy.

No seizures.

No metal in the head.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12
Dates: Start 1997-01; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] DeLong MR. Primate models of movement disorders of basal ganglia origin. Trends Neurosci. 1990 Jul;13(7):281-5. doi: 10.1016/0166-2236(90)90110-v. PMID 1695404
- [Background] Bergman H, Wichmann T, DeLong MR. Reversal of experimental parkinsonism by lesions of the subthalamic nucleus. Science. 1990 Sep 21;249(4975):1436-8. doi: 10.1126/science.2402638.
- [Background] Playford ED, Jenkins IH, Passingham RE, Nutt J, Frackowiak RS, Brooks DJ. Impaired mesial frontal and putamen activation in Parkinson's disease: a positron emission tomography study. Ann Neurol. 1992 Aug;32(2):151-61. doi: 10.1002/ana.410320206. PMID 1510355